CLINICAL TRIAL: NCT05005247
Title: A follow-on Study to Assess the Safety and Immunogenicity of a Booster Dose of GBS-NN/NN2 Vaccine 1 to 5 Years After GBS-NN/NN2 Recipients in Study MVX0002 Have Completed the Primary Vaccination Course, in Comparison With a Single Dose of GBS-NN/NN2 Administered in Placebo Participants From Study MVX0002 or Vaccine naïve Participants
Brief Title: Study to Assess a Booster Dose of GBS-NN/NN2 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minervax ApS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MVX0003
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Group B Streptococcus Infection

STUDY DESIGN:
Intervention Model Description: Open label booster vaccine study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GBS-NN/NN2 (Experimental): Single dose 0.5 millilitre (mL) intramuscular injection of GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS/NN2
  Interventions: Biological: GBS-NN/NN2

INTERVENTIONS:
Biological: GBS-NN/NN2 — GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS/NN2

SUMMARY:
This is an open label booster vaccine follow-up study. Participants who had received a primary course of GBS-NN/NN2 or placebo in Study MVX0002 will be invited to return to receive a booster dose (or first dose in the case of placebo or vaccine naïve participants) 1 to 5 years after the completion of the primary course of vaccination. All participants will receive a single dose of GBS-NN/NN2 containing 50μg of each fusion protein.

DETAILED DESCRIPTION:
This is an open label vaccine booster follow-up study. Participants who had received a primary course of GBS-NN/NN2 or placebo in Study MVX0002 will be invited to return to receive a booster dose (or first dose in the case of placebo or vaccine naïve participants) 1 to 5 years after the completion of the primary course of vaccination. All participants will receive a single dose of GBS-NN/NN2 containing 50μg of each fusion protein.

A minimum of 30 and a maximum of 40 female participants will be recruited, comprised of between 20 and 30 participants who had received previous vaccination with GBS-NN/NN2 in the MVX0002 study and up to 10 participants who had received placebo in the MVX0002 study. If an insufficient number of participants (less than 5) who previously received placebo return to this study, vaccine naïve participants will be recruited.

The study will include 7 visits: Visit 1 (Screening), Visit 2 (Day 1 dosing), Visit 3 (Day 8), Visit 4 (Day 29), Visit 5 (Day 57), Visit 6 (Day 85) and Visit 7 (Day 183 Follow-up).

ELIGIBILITY:
Inclusion Criteria:

To be confirmed at Screening:

1. Women who have participated in study MVX0002, with GBS-NN/NN2 vaccine and received active vaccine or placebo (unless it is necessary to recruit vaccine naïve participants to bolster the number of participants who received placebo in MVX0002).
2. Able to voluntarily provide written informed consent to participate in the study.
3. Healthy female participants aged 18-40 years (vaccine naïve participants only).
4. Female participant of childbearing potential willing to use a highly effective method of contraception (in addition to a condom for male partners), if applicable (unless of non-childbearing potential or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the participant) from the first dose until completion of the Day 85 visit. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. For the purposes of this study, this definition of a female of childbearing potential applies to all females in the study i.e., those who participated in the MVX0002 study and those who are considered vaccine naïve.
5. Female participant of non-childbearing potential. For the purposes of this study, this is defined as the participant being at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy).
6. Female participant with a negative pregnancy test at Screening and prior to dose.
7. Female participant of menopausal status confirmed by demonstrating at Screening that the serum level of the follicle stimulating hormone (FSH) falls within the respective pathology reference range. In the event a participant's menopausal status has been clearly established (for example, the participant indicates she has been amenorrhoeic for 10 years, confirmed by medical history, etc), but serum FSH levels are not consistent with a postmenopausal status, determination of the participant's eligibility to be included in the study will be at the Investigator's discretion following consultation with the Sponsor.
8. Body mass index (BMI) ≥18 and ≤30 kg/m2 (vaccine naïve participants only).
9. Participants' weight ≥ 50 kg and ≤ 100 kg at Screening (vaccine naïve participants only).
10. Non-smokers for at least 3 months prior to study vaccine administration.
11. No clinically significant abnormal test results for serum biochemistry, haematology and/or urine analyses within 28 days before dose administration of the IMP.
12. Participants with a negative urinary drugs of abuse (DOA) screen (including alcohol) test results, determined within 28 days before dose administration of the IMP (N.B.: A positive test result may be repeated at the Investigator's discretion, if on prescribed opiates resulting in a positive test, participants may be eligible at the investigators discretion).
13. No clinically significant abnormalities in vital signs (supine blood pressure/heart rate, respiration rate, tympanic temperature) determined within 28 days before dose of IMP.
14. Participants with a negative coronavirus (COVID-19) Reverse Transcription Polymerase Chain Reaction (RT-PCR) test on admission (Day 1 or Day-1 if deemed appropriate by the Principal Investigator (PI)) if required at the time.

To be re-confirmed prior to dose administration:

1. Participants continue to meet all screening inclusion criteria.
2. Participants with a negative urinary drugs of abuse screen (including alcohol) prior to dose administration.
3. Participants with a negative pregnancy test.
4. Participants with a negative COVID-19 RT-PCR test on admission (Day 1) (or Day -1 if deemed appropriate by the PI) if required at the time.

Exclusion Criteria:

To be confirmed at Screening:

1. Participants who have an autoimmune disease.
2. Participants who have a current infection or any significant illness at Screening (such participants can be rescreened once the active infection or significant illness has resolved).
3. Participants with history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, psychiatric, autoimmune disease or current infection.
4. Laboratory values at Screening which are deemed by the Investigator to be clinically significantly abnormal.
5. Positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab).
6. Participation in a clinical drug study during the 90 days or 5 half-lives, whichever is longer, preceding the initial dose in this study (such participants can be rescreened once the 90-day or 5 half-lives period has elapsed).
7. Participants with a history of severe allergic reactions after previous vaccination.
8. Participants with a history of hypersensitivity to the Investigational Medicinal Product (IMP) or any of the excipients within the IMP or documented allergy to aminoglycosides.
9. Participants who have received any vaccine within 7 days of dosing, or who are planning to receive a vaccine up to 7 days after receiving the GBS-NN/NN2 vaccine.
10. Participants who have received immunosuppressive therapy within the 6 months prior to Screening.
11. Participants with tattoos at the proposed site of vaccine administration.
12. Participants who, in the opinion of the Investigator, are unsuitable for participation in the study.
13. Pregnant or breast feeding.
14. Current or history of drug or alcohol abuse, or a positive urine alcohol test prior to dosing (prescribed opiates are acceptable).
15. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 28 days or 5 half-lives (whichever is longer) prior to the first dose of IMP with the exception of contraceptives and paracetamol (applies to vaccine naïve participants i.e., those who did not participate in the MVX0002 study and participants from the MVX0002 study (both active and placebo) who have not developed new medical conditions which require the use of chronic medications considered as permitted). If participants who participated in the MVX0002 study (either active or placebo recipients) have developed new medical conditions which require the use of chronic medications that do not affect the immune system, the inclusion of such participants will be permitted at the discretion of the Investigator on a case-by-case basis and, only if it is considered that the inclusion within the MVX0003 study will not be detrimental to participant safety.
16. Donation of blood or blood products within 90 days prior to vaccine administration.

To be re-confirmed prior to dose administration:

1. Development of any exclusion criteria since the Screening visit.
2. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements since the Screening visit with the exception of contraceptives and paracetamol (applies to vaccine naïve participants i.e., those who did not participate in the MVX0002 study and participants from the MVX0002 study (both active and placebo) who have not developed new medical conditions which require the use of chronic medications considered as permitted).
3. Participation in a clinical study since the Screening visit.
4. Donation of blood or blood products since the Screening visit.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Kitson, Study Director — gkitson@propharmapartners.uk.com
Locations (1):
- Simbec Clinical Pharmacology, Merthyr Tydfil, Wales, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on their participation on the previous MVX0002 study. The first participant was enrolled on August 17, 2021 and the last one was enrolled on August 8, 2022.
Pre-assignment Details: 27 patients were enrolled and received the study vaccine. 1 participant was withdrawn and not replaced (the participant requested withdrawal from the study).
Groups:
- MVX0002 25 μg GBS-NN/NN2: Patients received a booster dose of the group B streptococcus (GBS) vaccine GBS-NN/NN2 following an initial primary vaccination course with the vaccine GBS-NN/NN2 25 μg in the previous study MVX0002.
- MVX0002 50 μg GBS-NN/NN2: Patients received a booster dose of the group B streptococcus (GBS) vaccine GBS-NN/NN2 following an initial primary vaccination course with the vaccine GBS-NN/NN2 50 μg in the previous study MVX0002.
- MVX0002 Placebo/Vaccine Naïve: Vaccine naïve participants (either placebo recipients from study MVX0002 or new vaccine naïve participants) received a dose of the group B streptococcus (GBS) vaccine GBS-NN/NN2.
Period: Overall Study
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve
Started | 10 | 7 | 10
Completed | 10 | 6 | 10
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve | Total
Number analyzed (Participants) | 10 | 7 | 10 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 10 | 27
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.60) | 34.6 (5.83) | 29.2 (7.51) | 31.4 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 10 | 27
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 7 | 10 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 7 | 10 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 7 | 10 | 27
Height [Mean (Standard Deviation); unit: meters] | 1.644 (0.0578) | 1.639 (0.0805) | 1.633 (0.0691) | 1.639 (0.0658)
Weight [Mean (Standard Deviation); unit: kg] | 68.98 (6.870) | 68.33 (9.408) | 69.53 (9.625) | 69.01 (8.310)
BMI [Mean (Standard Deviation); unit: kg/m²] | 25.559 (2.6777) | 25.396 (2.3944) | 25.999 (2.4144) | 25.680 (2.4268)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Description: Number of participants with treatment emergent adverse events
Time Frame: 12 weeks (Day 85)
Measure: Count of Participants; unit: Participants
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve
Number analyzed (Participants) | 10 | 7 | 10
Participants
  Number of participants reporting at least one TEAE | 10 | 7 | 10
  Number of participants with Mild TEAE | 4 | 2 | 4
  Number of participants with Moderate TEAE | 6 | 5 | 6
  Number of participants with Severe TEAE | 0 | 0 | 0
  Number of participants with TEAE by relationship to Study Drug: Reasonable Possibility | 10 | 4 | 8
  Number of participants with TEAE by relationship to Study Drug: No Reasonable Possibility | 0 | 3 | 2

2. Secondary Outcome: Treatment Emergent Adverse Events
Description: Number of participants with treatment emergent adverse events
Time Frame: 6 months (Day 183)
Measure: Count of Participants; unit: Participants
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve
Number analyzed (Participants) | 10 | 7 | 10
Participants | 5 | 2 | 4

3. Secondary Outcome: Antibody Concentration Specific for GBS-NN and GBS-NN2 (Absolute Values)
Description: Absolute values of antibody concentration specific for GBS-NN and GBS-NN2
Time Frame: From Day 1 to Day 85
Population: Immunogenicity Set
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve
Number analyzed (Participants) | 10 | 6 | 10
μg/mL
  Anti-GBSNN antibodies : Day 1 (Absolute value) | 3.4314 [1.1644 to 10.1115] | 6.5606 [4.7386 to 9.0827] | 0.0838 [0.0363 to 0.1932]
  Anti-GBSNN antibodies : Day 85 (Absolute value) | 45.4768 [27.5667 to 75.0230] | 83.3289 [40.7246 to 170.5038] | 1.6497 [0.8161 to 3.3347]
  Anti-GBSNN2 antibodies : Day 1 (Absolute value) | 7.0260 [1.9392 to 25.4559] | 6.7734 [1.4783 to 31.0356] | 0.2275 [0.1365 to 0.3793]
  Anti-GBSNN2 antibodies : Day 85 (Absolute value) | 61.4636 [39.0362 to 96.7762] | 109.9307 [67.0156 to 180.3275] | 4.7237 [2.8023 to 7.9625]

4. Secondary Outcome: Antibody Concentration Specific for GBS-NN and GBS-NN2 (Fold Increase)
Description: Geometric mean fold increase in antibody concentration specific for GBS-NN and GBS-NN2
Time Frame: From Day 1 to Day 85
Population: Immunogenicity Set
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve
Number analyzed (Participants) | 10 | 6 | 10
ratio
  Anti-GBSNN antibodies (fold increase) | 13.25 [4.78 to 36.77] | 12.70 [6.32 to 25.52] | 19.70 [12.11 to 32.03]
  Anti-GBSNN2 antibodies (fold increase) | 8.75 [2.13 to 36.00] | 16.23 [4.49 to 58.61] | 20.76 [11.04 to 39.04]

5. Secondary Outcome: Antibody Concentration Specific for GBS-NN and GBS-NN2
Description: Geometric least square mean of antibody concentrations specific for GBS-NN and GBS-NN2 at day 85 of MVX002 study and day 1 and 85 of MVX003 study.
Time Frame: MVX002 day 85, MVX003 day 1 and MVX003 day 85
Population: Only participants who received placebo during the MVX0002 study were analyzed for this outcome measure in the "MVX0002 Placebo/Vaccine Naïve" arm. Vaccine naïve participants were excluded.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve
Number analyzed (Participants) | 10 | 6 | 5
μg/mL
  Anti-GBSNN Antibody - MVX002 Day 85 | 11.8 [4.37 to 31.7] | 22.6 [16.1 to 31.9] | 0.0247 [0.00426 to 0.144]
  Anti-GBSNN Antibody - MVX003 Day 1 | 3.43 [1.28 to 9.23] | 6.56 [4.66 to 9.24] | 0.0669 [0.0115 to 0.389]
  Anti-GBSNN Antibody - MVX003 Day 85 | 45.5 [22.1 to 93.6] | 83.3 [47.3 to 147] | 1.59 [0.396 to 6.40]
  Anti-GBSNN2 Antibody - MVX002 Day 85 | 29.1 [9.56 to 88.4] | 31.0 [8.57 to 112] | 0.117 [0.0411 to 0.330]
  Anti-GBSNN2 Antibody - MVX003 Day 1 | 7.03 [2.31 to 21.4] | 6.77 [1.87 to 24.5] | 0.206 [0.0726 to 0.584]
  Anti-GBSNN2 Antibody - MVX003 Day 85 | 61.5 [30.1 to 126] | 110 [50.1 to 241] | 4.42 [1.52 to 12.8]

ADVERSE EVENTS:
Time Frame: From screening to end of safety follow-up.
Description: All Adverse Events (AEs) were recorded, whether considered minor or serious, drug-related, or not.
  From vaccination (Day 1) to Day 7 solicited and unsolicited AEs were recorded. The following AE were solicited : Injection site reactions, fatigue, headache, myalgia and Influenza like illness.
  From Day 8 to Day 85 only unsolicited AEs were collected. From Day 86 to Day 183 all AEs were recorded in the Patient Diary Card and evaluated at Visit 7.
Arm/Group | MVX0002 25 μg GBS-NN/NN2 | MVX0002 50 μg GBS-NN/NN2 | MVX0002 Placebo/Vaccine Naïve
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 7/7 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVX0002 25 μg GBS-NN/NN2 (N=10) | MVX0002 50 μg GBS-NN/NN2 (N=7) | MVX0002 Placebo/Vaccine Naïve (N=10)
Injection site reaction (General disorders) | 10 (10) | 6 (6) | 8 (8) — Pain, redness, bruising, tenderness, itching and swelling.
Headache (Nervous system disorders) | 6 (13) | 3 (5) | 8 (13)
Fatigue (General disorders) | 5 (5) | 2 (2) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 5 (5)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic fatigue syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (2)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05005247/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT05005247/SAP_001.pdf